CLINICAL TRIAL: NCT03857984
Title: Hemodialysis and Erythrocyte Fatty-Acid Status: a Lipidomics Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin Gollasch (Other)
Responsible Party: Sponsor-Investigator, Benjamin Gollasch, Principal Investigator, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E2/113/08
Record Dates: First submitted 2019-02-24; First posted 2019-02-28 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Fatty Acid Metabolism; Erythrocytes; Lipidomics; Hemodialysis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Erythrocyte Fatty-Acid Status (Experimental): Erythrocyte Fatty-Acid Status Profiling of HD patients are studied before and after a single HD using LC-MS / MS
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — blood sample before and after a single HD

SUMMARY:
Hypotension with potentially serious consequences for organ perfusion is a common complication in extracorporeal procedures such as hemodialysis / hemofiltration. The exact reasons for this are still insufficiently clarified. Probably periinterventional vasorelaxant released substances play a crucial role in these procedures. These substances could be due to contact of blood cells with the Membrane in the dialyzer / hemofilter arise. In this project the hypothesis will be checked, if EETs / DHETs are released by Erythrocytes during hemodialysis and thus act as potential candidate products for the result of hypotonic phases in the Dialysis.

We will determine differences in RBC fatty acids profiling in hemodialysis patients before and after dialysis intervention. Furthermore a matched control group of healthy individuals will be profiled. RBC fatty acids profiling will be achieved by using targeted HPLC-MS mass spectrometry.

It is believed that during hemodialysis / HLM / CVVH there is an increase in EETs / DHETs in the serum and in the erythrocytes. It is believed that shear forces play an important role in the release of erythrocyte EETs / DHETs.

DETAILED DESCRIPTION:
Differences in Erythrocyte Fatty-Acid Status Profiling in:

* before and after hemodialysis intervention
* in hemodialysis patients and healthy individuals Venous blood will be collected from each subject in the sitting position

ELIGIBILITY:
Inclusion Criteria for hemodialysis patients:

* Patients who have a history of renal failure and undergo hemodialysis / hemofiltration
* Age over 18 years
* Ability to consent
* There is a written consent of the study participant

Exclusion Criteria for healthy control group:

* chronic illness requiring any medication
* pregnancy
* limitations regarding functioning in the hypoxic chamber
* inability to follow simple instructions relevant or severe abnormalities in medical history, physical examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation of relative quantities of erythrocyte fatty-acid parameters related to its dynamic during Hemodialysis, using LC-MS / MS. | 4-5 Months
  EETs / DHETs will be analyzed in the erythrocytes and serum of the recovered blood samples.
  The determination will made in cooperation with a Berliner Biotech company. This involves liquid chromatography with MS coupling (LC-MS / MS) used. The data analysis is carried out by means of suitable statistical methods to perform erythrocyte fatty-acid status profiling.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Experimental & Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided